CLINICAL TRIAL: NCT04100421
Title: Study on the Level of Bisphenol Compounds in Patients With Chronic Kidney Disease and Renal Replacement Therapy and Relationship Between Bisphenols and Dialyzer Membrane
Brief Title: Exposure Of Bisphenol Analogues In Chronic Kidney Disease and Dialysis Patients
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Ding Feng, Kidney internal medicine professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: BPs
Record Dates: First submitted 2019-09-21; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Diseases; Hemodialysis Complication
Keywords: bisphenol; human exposure; chronic kidney disease; blood purification
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Mild renal injury: CKD patients with eGFR ≥ 60 ml∙min-1∙ (1.73 m2)-1. The eGFR was evaluated by the Chronic Kidney Disease Epidemiology Collaboration (eGFR-EPI).
- Moderate renal injury: CKD patients with eGFR between 30 ml∙min-1∙(1.73 m2)-1 to 60 ml∙min-1∙(1.73 m2)-1. The eGFR was evaluated by the Chronic Kidney Disease Epidemiology Collaboration (eGFR-EPI).
- Severe renal injury: CKD patients with eGFR < 30 ml∙min-1∙(1.73 m2)-1. The eGFR was evaluated by the Chronic Kidney Disease Epidemiology Collaboration (eGFR-EPI).
- Hemodialysis: uremic patients on hemodialysis therapy
- Peritoneal dialysis: uremic patients on peritoneal dialysis
- Healthy control: Healthy volunteers with no history of kidney diseases or any chronic diseases which may lead to renal injury.

SUMMARY:
In this retrospective study, the serum levels of Bisphenol A (BPA) and three BPA analogs, namely, bisphenol B (BPB), bisphenol S (BPS), and bisphenol F (BPF), in patients with CKD, patients on dialysis therapy and healthy control were investigated to find out if BPA and BPA analogs accumulates in patients with chronic kidney disease (CKD), and if hemodialysis filters contribute to bisphenol burden in patients on hemodialysis (HD).

ELIGIBILITY:
Inclusion Criteria:

* age 18; informed consent

Exclusion Criteria:

* absence of active inflammatory, infectious, malignant diseases, acute chronic kidney disease, or pregnancy at the initiation or during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with CKD, on dialysis in one center, and age- and gender- matched healthy volunteers were enrolled from Shanghai Ninth People's Hospital affiliated to Shanghai JiaoTong University.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Death | 2017.01-2018.06

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, China